CLINICAL TRIAL: NCT02450214
Title: Efficacy of Ketamine and Magnesium Association in the Postoperative Pain After Liposuction and Lipoabdominoplasty: Prospective, Randomized and Blinded Study
Brief Title: Intraoperative Ketamine and Magnesium Therapy for Control of Postoperative Pain After a Liposuction and Lipoabdominoplasty
Acronym: KEMPLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Veronica Varas Vega, MD, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OAIC N 722/15
Record Dates: First submitted 2015-05-18; First posted 2015-05-21 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2016-10

CONDITIONS: Pain, Postoperative
Keywords: Ketamine; Magnesium; Analgesia; Liposuction; Lipoabdominoplasty; Preemptive analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Sodium Chloride; Ketamine; Magnesium

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Control group (C) (Sham Comparator): 50 mL syringe with saline, plus 1 flask of 100 mL saline (Saline)
  Interventions: Drug: Saline
- Ketamine group (K) (Experimental): 50 mL syringe with ketamine (50mg / 50ml), plus 1 flask of 100 mL saline (Ketamine)
  Interventions: Drug: Ketamine
- Magnesium + ketamine group (MGK) (Experimental): 50mL syringe with ketamine (50mg / 50ml), plus a flask of 100ml of saline with 5 g of magnesium sulfate (Ketamine + magnesium)
  Interventions: Drug: Ketamine + magnesium

INTERVENTIONS:
Drug: Saline — 50 mL syringe will be infused at 0.3 mL/Kg in bolus and then 0.15 mL/Kg/h 100 mL flask will be infused at 1mL/Kg in bolus for 30 min and then 0.25mL/Kg/h
  Arms: Control group (C)
Drug: Ketamine — 50 mL syringe will be infused at 0.3 mL/Kg in bolus and then 0.15 mL/Kg/h 100 mL flask will be infused at 1mL/Kg in bolus for 30 min and then 0.25mL/Kg/h
  Arms: Ketamine group (K)
Drug: Ketamine + magnesium — 50 mL syringe will be infused at 0.3 mL/Kg in bolus and then 0.15 mL/Kg/h 100 mL flask will be infused at 1mL/Kg in bolus for 30 min and then 0.25mL/Kg/h
  Arms: Magnesium + ketamine group (MGK)

SUMMARY:
Lipoabdominoplasty and liposuction are one of the most common plastic surgeries. The management of postoperative pain is complex. Non Steroidal Anti Inflammatory Drugs (NSAIDs) are insufficient, while opioids are avoided by their adverse effects and regional techniques are hampered by a premature discharge. In this context, the investigators seek an intraoperative multimodal analgesic technique blocking NMDA receptors with ketamine plus magnesium to significantly decrease postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Female and male
* 18 years or older
* Liposuction and lipoabdominoplasty
* ASA 1 and 2
* BMI 21-28 Kg/m2
* Full secondary education

Exclusion Criteria:

* Patients with surgeries added to the main proceedings
* Scheduled to tuck in Flor de Lis or Body Lift
* History of use of analgesic drugs 48 hours before surgery
* Peripheral central neurological diseases
* Known allergy will be excluded to medication in use in this study (ketamine, magnesium, clindamycin and penicillin or other)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-06; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Opioids consumption | 12 h after surgery
Postoperative Pain (Postoperative Pain and Disability Scale) | 2, 7, 14, 21, 45 and 90 days after surgery
  Postoperative Pain and Disability Scale (Body-PPDS) will be used to quantify pain

SECONDARY OUTCOMES:
Early postoperative pain (Visual analogue pain scale) | 0, 2, 4, 6, 12 and 24 h after surgery
  Visual analogue pain scale (0-10) will be used to quantify pain
Early postoperative pain (Time to first request for supplemental analgesia) | 1 day
  Time to first request for supplemental analgesia.
Disability (Time delay in returning to work) | 90 days
  Time delay in returning to work.
Postoperative Chronic Pain (McGill scale) | Day after surgery, 7, 30 and 90 days after surgery
  McGill scale for chronic painwill be used to quantify pain

OTHER OUTCOMES:
Drug Side Effect | First day after surgery
  Hallucinations, unpleasent dreams or some patient discomfort, sedation level, pruritus, hypotension, bradycardia, urinary retention, nausea, vomiting.
Other Variables | First day
  Sociodemographic variables; surgical variables as liters of aspirated fat, weight of resected flap, operative time, bleeding measured as the difference between pre and postoperative hemoblobinemia, immediate postoperative complications such as bleeding or hematoma and thromboembolic complications; anesthetic variables as total amount of remifentanil and sevorane consumption.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico de la Universidad de Chile, Santiago, RM, Chile